CLINICAL TRIAL: NCT02521220
Title: Beneficial Effects of the Amino-acid Food Supplement L-citrulline in Participants With Peripheral Artery Disease
Brief Title: L-Citrulline in Peripheral Artery Disease
Acronym: CIPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Clinical Trial Center Maastricht B.V. (Other); Catharina Ziekenhuis Eindhoven (Other); Hannover Medical School (Other)
Responsible Party: Principal Investigator, H. Schmidt, Prof., Maastricht University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIPER2015UM
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Peripheral Arterial Disease
Keywords: L-citrulline; Endothelial dysfunction
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-citrulline (Experimental): Oral food-supplemental amino-acid L-citrulline. 2 times 3g per day.
  Interventions: Dietary Supplement: L-citrulline
- Maltodextrin (Placebo Comparator): Maltodextrin as placebo. 2 times 3g per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-citrulline — L-citrulline 2 times daily 3 gram (6g/day)
  Arms: L-citrulline
Dietary Supplement: Placebo — Maltodextrin 2 times daily 3 gram (6g/day)
  Arms: Maltodextrin

SUMMARY:
Some studies have reported improved vascular function with the supplementation of L-arginine in participants with cardiovascular disease (CVD). Several clinical studies have also begun the investigation of L-arginine supplementation in participants with peripheral artery disease (PAD). This is particularly important as currently there are limited options available to medically manage intermittent leg pain resulted from PAD. Although some of these short-term clinical trials suggested that oral L-arginine improved walking distance or improved walking speed in participants with PAD, these results were not consistent. Further, only 1% of the oral supplemented L-arginine is available for the NO production as the rest is metabolised by the body. A better way to provide the body with substrate to produce NO is therefore needed. The natural amino acid and food component, L-citrulline has been suggested to be a good candidate for this purpose.

L-citrulline, named after watermelon citrullus vulgaris from which it was first isolated, is a natural precursor of L-arginine. Studies have shown that L-citrulline is metabolised by the body to a lesser degree compared to L-arginine and hence is an effective precursor of arginine in peripheral tissues, including endothelial cells. Oral L-citrulline supplementation also eliminates some of the unwanted effects associated with oral arginine supplementation and it is well tolerated without known side effects. In addition, L-citrulline is a supplement that is available over-the-counter. Thus, oral supplementation of L-citrulline may be a new intervention strategy in participants with PAD.

The investigators hypothesize that the oral food supplement L-citrulline, unlike L-arginine, reverses endothelial dysfunction. In a multinational, multicenter, double blinded, randomised, placebo-controlled cross-over trial the effects of L-citrulline in peripheral artery disease will be investigated.

DETAILED DESCRIPTION:
The primary aim of this trial is to examine whether the oral food supplement L-citrulline has any effect on clinical status, walking distance, arterial and endothelial function in participants with PAD.

The investigators will use a double-blinded crossover design in which patients serve as their own controls. Patients who are enrolled will have two 'treatment' periods of twelve weeks with a wash-out period of 4 weeks in between. Patients will be randomly assigned to get L-citrulline in the first and placebo in the second period and vice versa.

After a screening phase of 3 weeks, there will be a 'zero-point' measurement en then the first 'treatment' period of 12 weeks starts (placebo or food-supplement). Then there is a wash-out phase of 4 weeks after which the second 'treatment' period starts (food-supplement or placebo) In both periods, after 2 weeks and at the end of the period, a measurement of primary and secondary outcomes will be done: a questionnaire has to be filled out, treadmill test and flow-mediated dilation (for vessel function). The follow-up will take another 4 weeks and will end with a phone call to check for the condition of the patient and possible side effects.

Since every patient gets both placebo and the food-supplement, every patient is his/her own control.

The study was completed with 24 patients in Hannover, Germany, and 25 in Melbourne, Australia.

ELIGIBILITY:
Inclusion Criteria:

* 40 years or older males and postmenopausal women;
* male participants must agree to using an adequate form of contraception during the study period;
* 6-month history of stable intermittent claudication (IC) due to PAD;
* PAD secondary to atherosclerosis with significant claudication (Fontaine class II defined as IC, or Fontaine class III defined as pain at rest);
* IC characterised by pain, ache, cramp, numbness or severe fatigue involving muscles of one or both lower extremities, reproducibly provoked by walking and relieved by rest;
* ankle-brachial index (ABI) at rest of <0.9 and at least 25% decrease in ABI within 1 min during exercise recovery;
* capacity to walk more than 2 min/15 meters but no more than 12 min on a treadmill using the Skinner-Gardner protocol;
* walking limited by claudication, not coexisting conditions; and
* difference between two consecutive baseline exercise treadmill tests of <25% during the 3-weeks run-in period; and
* no change in medications or physical activity within 3 months prior to enrolment.

Exclusion Criteria:

* Women of child-bearing potential;
* Current enrolment in another clinical trial and/or ingestion of another investigational product within the past 30 days before enrolment;
* PAD of non-atherosclerotic nature;
* Fontaine class IV i.e. ulcer or gangrene;
* leg amputation above the ankle;
* peripheral vascular surgery, sympathectomy, peripheral angioplasty or stent insertion within the previous 3 months;
* myocardial infarction, unstable angina, percutaneous transluminal coronary angioplasty or coronary artery bypass graft surgery within the previous 3 months;
* uncontrolled hypertension (resting systolic blood pressure (SBP) >190 or diastolic blood pressure (DBP) >115 mmHg);
* hypotension (SBP <90mmHg);
* type I diabetes, proliferative retinopathy;
* history of disease state or surgery that affects gastrointestinal absorption;
* significant renal disease (serum creatinine >3.0 mg/dl);
* liver disease (transaminase > 3x upper limit of normal, bilirubin >1.5 times upper limits of normal);
* history of treatment for any malignancy within the past 5 years, or evidence of active malignancy other than squamous cells or basal cell carcinoma of the skin;
* serious infection or hypotension associated with sepsis in the last month;
* cerebrovascular infarct in the last 3 months;
* autoimmune disorders (e.g. systemic lupus erythematosis, ulcerative colitis);
* any other acute or chronic medical condition that in the opinion of the investigators increases the likelihood that the participant would be unable to complete the study;
* unwillingness to discontinue arginine- or L-citrulline-containing products, pentoxifylline, L-carnitine, or prostacyclin for at least 1 month prior to and during the study; and
* conditions other than PAD that limit walking distance.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Absolute claudication distance | 30 weeks
  Measurement of absolute claudication distance using a treadmill exercise test

SECONDARY OUTCOMES:
Endothelial function using endo-PAT (peripheral arterial tone) | 30 weeks
  Flow mediated dilation

OTHER OUTCOMES:
L-citrulline metabolites | 30 weeks
  Blood plasma levels of L-citrulline, L-arginine and asymmetric dimethylarginine (ADMA)
Walking impairment questionnaire | 30 weeks
  Assessment of functionality with regard to walking using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Harald Schmidt, Prof., Principal Investigator — Maastricht University
Locations (3):
- Hannover Medical School, Hanover, Germany
- Netherlands (2):
  - Maastricht University, Maastricht, Limburg
  - Catharina Ziekenhuis Eindhoven, Eindhoven

IPD SHARING:
Plan to Share IPD: Undecided